CLINICAL TRIAL: NCT06262048
Title: Prevention of Post Operative Urinary Retention After Thoracic Surgery: A Phase II Feasbility Trial
Brief Title: Prevention of Post Operative Urinary Retention After Thoracic Surgery Trial
Acronym: PrePOURTS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Rahul Nayak, MD MSc FRCSC, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PrePOURTS
Record Dates: First submitted 2024-01-15; First posted 2024-02-15 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Urinary Retention Postoperative
Keywords: urinary retention; thoracic surgery; urinary catheter
MeSH Terms: conditions — Urinary Retention | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: single centre, double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Tamsulosin
  Interventions: Drug: Tamsulosin Hydrochloride
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tamsulosin Hydrochloride — 2 days pre-op, day of surgery, 2 days post-op
  Other Names: tamsulosin HCL
  Arms: Treatment
Other: Placebo — 2 days pre-op, day of surgery, 2 days post-op
  Arms: Placebo

SUMMARY:
The objectives of this study are to determine the feasibility of conducting a full-scale randomized control trial comparing the efficacy of tamsulosin compared to placebo in reducing post-operative urinary retention in people undergoing elective thoracic surgery.

DETAILED DESCRIPTION:
The objectives of this study are to determine the feasibility of conducting a full-scale randomized control trial comparing the efficacy of tamsulosin compared to placebo in reducing post-operative urinary retention in people undergoing elective thoracic surgery. Primary outcomes being measured are the enrollment rate, protocol adherence rate and participant drop out.

ELIGIBILITY:
Inclusion Criteria ( 2 or more of the following risk factors):

* Male Sex
* Age greater than or equal to 40 years
* History of Diabetes Mellitus
* Prior pelvic irradiation
* Use of indwelling Thoracic Epidural analgesia
* Prior history of urinary retention

AND

International Prostate Specific Score greater than or equal to 1.

Exclusion Criteria:

* Active treatment of Benign Prostatic Hyperplasia (BPH)
* Hypersensitivity or allergy to tamsulosin HCL
* Active treatment with tamsulosin or other alpha-blocker or uses of tamsulosin/ other alpha-blocker within 3 weeks of enrollment date
* Active urinary tract infection
* History of urological disorder specified as urethral stricture, BPH, bladder or prostate malignancy.
* History of urological surgery (Transurethral resection of the Prostate, Transurethral resection of the Bladder, Bladder suspension, prostatectomy)
* Underlying neurological disorders resulting in impaired bladder function
* Any known contraindication to the use of tamsulosin HCL
* Nursing/ Breastfeeding women
* Use of intraoperative bladder catheter
* patients for whom cataract and/or glaucoma surgery is scheduled.
* patients on strong inhibitors of CYP3A4 (e.g., ketoconazole), on moderate inhibitors of CYP3A4 (e.g., erythromycin), on strong (e.g. paroxetine), on moderate (e.g., terbinafine) inhibitors of CYP2D6 or in patients known to be CYP2D6 poor metabolizers.
* patients with a serious or life-threatening sulfa allergy
* patients with severe hepatic insufficiency
* patients with severe renal impairment (creatinine clearance of <10 mL/min)
* patients with a serious or life-threatening sulfa allergy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment Effectiveness | 4 months
  Percentage of Screen eligible patients consenting to the study
Monthly recruitment | 4 months
  Rate of monthly recruitment
Protocol adherence | 4 Months
  Percentage of enrolled patient adherent to protocol during intervention phase

SECONDARY OUTCOMES:
Rate of Straight Catheterizations | 30 days post-op
  Number of Single urinary catheterizations performed
Rate of Indwelling Catheterizations | 30 days post-op
  Proportion of patients who have an indwelling foley catheter inserted during their post-operative stay
Time to first catheterization | up to 30 days post-op
  Time to first catheterization
Treatment Related Adverse Events | 30 days post-op
  Unexpected or noxious events that occur as a result of or suspected to be a result of use of the study drug.
Catheter related complications | 30 days post-op
  Rates of catheter related complications within 30 days of catheterization (e.g. CAUTI, Urethral Trauma, Hematuria, urethral stricture)
Length of stay | 30 days post-op
  Duration of hospital length of stay will be measured by collecting the date of admission and the date of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Nayal, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No